CLINICAL TRIAL: NCT06871943
Title: Developing a Rationale for the Use of Breathing Frequency and Wearable Foot-pods to Measure Intensity in Cardiac Populations
Brief Title: Can Wearable Technology be Used to Predict Exercise Intensity
Acronym: (CWTPEI)
Status: Not yet recruiting | Type: Observational
Sponsor: Keele University (Other)
Collaborators: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KeeleU; RG-0393-24 (Other: Integrated Research Application System)
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction (MI)
Keywords: aerobic capacity; breathing frequency; walking capacity
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myocardial Infraction: Participants who have suffered a myocardial infraction in the past 6 months and are actively enrolled onto a cardiac rehabilitation programme
  Interventions: Other: Incremental Shuttle Walk Tests

INTERVENTIONS:
Other: Incremental Shuttle Walk Tests — The participants will walk on the flat around cones placed 9 meters apart inline with the procedure for the incremental shuttle walk test. They will also walk at a matched speed to the incremental shuttle walk test on a treadmill. This will be performed in a counter balanced procedure to reduce any benefit of a learning effect.
  Other Names: ISWT

SUMMARY:
There is a knowledge gap in the literature around using watts to measure exercise intensity in walking and running, this is largely due to new technological developments. Whereas the relationship is widely recognised and used for cycling in elite to clinical populations.

While the relationship breathing rate and exercise intensity is well established, this are no guidelines using breathing rate as a physiological measure of intensity. New technology may aid to bridge these gaps.

The main aims of the study are: -

Can the relationship between oxygen uptake and watts during incremental exercise Can breathing frequency be used to determine aerobic exercise intensity

The participants will complete two 9 minute incremental accredited exercise tests on the flat around cones and on treadmill at the given speed of walking around the cones. The test will stop at 6.8kph or at participant volition.

DETAILED DESCRIPTION:
The experimental feasibility study involves testing if the wearable technology (Stryd accelerometer) can translate work rate into an accurate measurement of watts (energy produced) within cardiac populations, when compared to V̇o2 consumed. While also testing to see the measured relationship between breathing rate and exercise induced exertion levels. The testing will involve participants working to a sub maximal incremental shuttle walk test pace on treadmill (unto 6.8kph) and following standard procedure on the flat around cones. They will be wearing a Stryd accelerometer attached to their training shoes and Respa breathing monitor attached to their lapel or t-shirt. V̇o2 will be measured using a Cortex Metalyzer 3B. All participants will perform the testing twice in a counter balanced order (i.e participant one will perform the treadmill first, while the next will perform the testing on the flat around cones).

Participants will be recruited from the cardiac rehabilitation team at the University Hospital of the North Midlands.

The pace of the treadmill will be in line with the constant walking pace required to achieve a steady state at each level of the incremental shuttle walk test protocol. The treadmill will not be an incline as normal testing is on flat surface. The Stryd and Respa will be linked to a mobile device where watts and breathing frequency readings will be gathered, progression to the next stage will be at one minute.

Each test lasts for 9 minutes, with a 15-minute recovery period between tests and pre and post exercise tests, participation will take approximately 1 hour. Post testing the participant can remove the device and face mask; while being encouraged to cool down until heart rate is within 20 beats of resting levels but they can leave at any time.

Power will be measured in watts from the Stryd accelerometer, V̇O2 will be measured in ml.kg.min, while respiratory rate will be breaths per minute To remove anomalies from the excel sheet, the watts and breathing frequency readings will be taken from smoothing the data within the last 30 seconds of the level. This will allow the participant to adjust to the change in pace and achieve a steady state of walking. The V̇o2 reading will also be taken in the last 30 seconds with the average of the smoothed data used.

It is anticipated that all participants will not finish the testing up to stage 9, due to volitional fatigue. All data will be reported and recorded, with a n value for each stage, denoting the power and the perceived drop out at each point.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial Infraction in the past 6 months
* Able to walk on a treadmill
* Aged ≥ 18

Exclusion Criteria:

• Injury or condition that impedes normal gait

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have suffered an myocardial infraction in the last 6 months and be actively participating in the cardiac rehabilitation programme at the University Hospital of North Midlands in the United Kingdom
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Can a Stryd accelerometer be used to predict V̇o2max and therefore be used to gather a baseline for exercise prescription in cardiac populations post myocardial infraction. | 1 day of testing, enrolment may be within 1 month prior to the test
  Develop a regression equation for the use of watts derived from a foot pod to predict vo2. Assessing watts per kg of body mass against vo2 per kg of body mass, offering insight as to how this population group can use watts to prescribe exercise.

SECONDARY OUTCOMES:
Can a breathing frequency monitor be used to predict aerobic exercise intensity in cardiac populations post myocardial infraction. | 1 day of testing, enrolment may be within 1 month prior to the test
  Develop a regression equation for the use of breathing frequency to predict vo2. Assessing breathing frequency against vo2 per kg of body mass, offering insight as to how this population group can use watts to prescribe exercise.

CONTACTS AND LOCATIONS:
Overall Officials: John Buckley, PhD, Study Chair — Keele University

IPD SHARING:
Plan to Share IPD: Undecided
Further studies may be shared but this stage of the research process is too earlier.

REFERENCES:
- See also: Page 220 details a conference abstract from the European Congress for Sports Science at which an initial study on healthy participants was presented — https://www.ecss.mobi/DATA/CONGRESSES/GLASGOW_2024/DOCUMENTS/2024_BOA_Web.pdf